CLINICAL TRIAL: NCT02683096
Title: Screening for Congenital Cytomegalovirus Infection in Newborns With Failed Hearing Screen or Who Are Small for Gestational Age
Brief Title: Screening for Congenital Cytomegalovirus Infection in Newborns
Acronym: CMV
Status: Completed | Type: Observational
Sponsor: Southern Illinois University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: ROD-SIU-15-288-CMV
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva PCR assays
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SGA Infants
  Interventions: Other: Observation
- Failed Hearing Screen Infants
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Viable Infants with a failed hearing screen or a diagnosis of SGA who are born at either St. John's Hospital or MMC at ≥ 28 weeks gestation.

SUMMARY:
Our central hypothesis is that screening newborn infants who either fail their newborn hearing test or have a diagnosis of small for gestational age (SGA) will lead to better identification of infants with congenital CMV infection and enhanced rates of therapeutic intervention. This has the potential to significantly improve outcomes for infants with this common viral infection. This particular cohort of patients have not been well studied locally or regionally. In addition, in view of current legislation that will be effective in January, 2016 this is a timely project that will provide preliminary data for future statewide recommendations around CMV testing of newborn infants. This will be a pilot/feasibility study to obtain preliminary data for an Illinois Department of Public Health (IDPH) Title V grant. Although not guaranteed, preliminary discussions with the IDPH are highly encouraging giving the statewide interest in this topic.

DETAILED DESCRIPTION:
Congenital cytomegalovirus (CMV) infection is the leading non-genetic cause of sensorineural hearing loss (SNHL) in children in the United States, and is the most frequent known viral cause of mental disability. Approximately one percent of all newborn infants in the United States are infected with CMV. Of those infected, approximately 10% have involvement that is evident at birth (symptomatic congenital CMV disease) with manifestations including microcephaly, central nervous system abnormalities, chorioretinitis, hepatosplenomegaly, and SNHL. The most common sequelae following congenital CMV infection is SNHL and it occurs in up to 50% of infants with symptomatic congenital CMV infection and in 15% of asymptomatic infants. Overall, congenital CMV infection accounts for one-third of all cases of SNHL. Among newborn infants who fail hearing screening, the prevalence of congenital CMV infection is much higher (six to 10%) than the general newborn population (<1%). Since early therapeutic intervention for infants with symptomatic congenital CMV infections improves audiological and neurodevelopmental outcomes early diagnosis is essential for early treatment and maximizing infant outcomes.

The Illinois Legislature passed a bill that was signed into law in August 2015 by Governor Rauner regarding congenital CMV. The main objectives of this law are public education regarding CMV infection and efforts to raise awareness of this infection amongst healthcare providers caring for expectant mothers. This Public Act mandates parents receive information regarding testing opportunities and early intervention services for CMV infection when their newborn infant fails his or her hearing screen. Although this bill does not mandate CMV screening, it does state that the hospitals have to provide information about testing options.

Our central hypothesis is that screening newborn infants who either fail their newborn hearing test or have a diagnosis of small for gestational age (SGA) will lead to better identification of infants with congenital CMV infection and enhanced rates of therapeutic intervention. This has the potential to significantly improve outcomes for infants with this common viral infection. This particular cohort of patients have not been well studied locally or regionally. In addition, in view of current legislation that will be effective in January, 2016 this is a timely project that will provide preliminary data for future statewide recommendations around CMV testing of newborn infants. This will be a pilot/feasibility study to obtain preliminary data for an Illinois Department of Public Health (IDPH) Title V grant. Although not guaranteed, preliminary discussions with the IDPH are highly encouraging giving the statewide interest in this topic.

ELIGIBILITY:
Inclusion Criteria:

* Viable Infants with a failed hearing screen or a diagnosis of SGA who are born at either St. John's Hospital or MMC at ≥ 28 weeks gestation.

Exclusion Criteria:

* Infants born ≤ 27 weeks gestation, infants who are not SGA, infants who pass their newborn hearing screen.

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants who either fail their newborn hearing test or have a diagnosis of small for gestational age (SGA)
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Measure the incidence of congenital CMV infection in neonates with failed hearing screen. | At birth
Measure the incidence of congenital CMV infection in neonates who are SGA. | At birth

SECONDARY OUTCOMES:
Measure the proportion of patients that receive therapeutic intervention in 2 groups of patients with congenital CMV infection | First six months of life

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Rodriguez, MD, Principal Investigator — SIU School of Medicine

IPD SHARING:
Plan to Share IPD: No